CLINICAL TRIAL: NCT07132229
Title: Impact of Cervical High-Intensity Resistive Exercises on Ventilatory Measures in Patients With Chronic Non-Specific Neck Pain
Brief Title: Impact Of Cervical High-Intensity Resistive Exercises In Patients With Chronic Non-Specific Neck Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Taha Ahmed Taha Elbragily, PhD Candidate in Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004930
Record Dates: First submitted 2025-08-05; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Chronic Non-specific Neck Pain
Keywords: neck pain; cervical pain; High-Intensity Resistive Exercises
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical High-Intensity Resistive Exercises + Conventional physical therapy (Experimental): Patients in this group will receive Cervical High-Intensity Resistive Exercises + Conventional physical therapy
  Interventions: Other: Cervical High-Intensity Resistive Exercises; Other: Conventional physical therapy
- Conventional physical therapy (Active Comparator): Patients in this group will receive Conventional physical therapy
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Cervical High-Intensity Resistive Exercises — The patient will wear a neck harness, and a weight equivalent to 90% of the patient's measured maximum voluntary isometric contraction (MVIC) will be attached to it.
  Arms: Cervical High-Intensity Resistive Exercises + Conventional physical therapy
Other: Conventional physical therapy — Conventional physical therapy consisting of TENS for pain control, soft tissue release for the cervical and associated muscles, activation and strengthening exercises for the deep neck flexors, extensors, and scapular muscles, as well as diaphragmatic breathing exercises.

SUMMARY:
Purposes of the study

To investigate the effect of adding Cervical High-Intensity Resistive Exercises to conventional physical therapy in patients with Chronic Non-Specific Neck Pain

DETAILED DESCRIPTION:
Patients will be randomized into either Cervical High-Intensity Resistive Exercises group or Conventional physical therapy group. Patients will receive the intervention for six weeks. Outcomes will be assessed at baseline and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Thirty-four patients diagnosed CNSNP.
2. Age of the patients between 20-40 years.
3. Non-specific neck pain started more than 3 months.
4. Reduce ventilatory function; FVC >= 70% from predicted.
5. Waist to height ratio (WtHR)> 60 %.
6. Positive craniocervical flexion test.
7. Positive neck flexor endurance test.
8. Pain at neck after prolonged static weight bearing positions.
9. Pain with palpation of the neck paraspinal or suboccipital or trapezius muscles.

Exclusion Criteria:

1. History of whiplash injury.
2. Clinical sign of cervical radiculopathy.
3. Clinical signs of cervical myelopathy.
4. Rheumatoid Arthritis or any other autoimmune diseases.
5. Any respiratory disorders.
6. Tumors.
7. vertebrobasilar insufficiency VBI.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Disability | Change from Baseline Disability at 6 weeks
  Neck disability index (NDI)
Diaphragm thickness | Change from Baseline Diaphragm thickness at 6 weeks
  Ultrasound
Forced vital capacity (FVC) | Change from Baseline Forced vital capacity (FVC) at 6 weeks
  Spirometry
maximum voluntary ventilation (MVV) | Change from maximum voluntary ventilation (MVV) at 6 weeks
  Spirometry

SECONDARY OUTCOMES:
Neck pain | Change from Baseline Neck pain at 6 weeks
  Visual analogue scale
Strength of neck flexors, extensors, and side bending | Change from Baseline Strength of neck flexors, extensors, and side bending at 6 weeks
  Hand-held dynamometer (HHD)

CONTACTS AND LOCATIONS:
Locations (1):
- outpatient clinic, Faculty of Physical Therapy, Cairo University, Giza, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Undecided